CLINICAL TRIAL: NCT02783872
Title: Neurodevelopmental Substrates of Emotion Regulation in Overweight, Binge Eating Youth
Brief Title: Emotion Regulation and Binge Eating in Youth With Obesity
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Miriam H
Record Dates: First submitted 2016-05-20; First posted 2016-05-26 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Binge-Eating Disorder
MeSH Terms: conditions — Obesity; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Loss of control: 30 overweight or obese (BMI≥85th %ile) youth endorsing loss of control eating within the past 3 months
- Overweight control: 30 overweight or obese controls without any history of loss of control eating
- Normal-weight control: 15 normal-weight controls without any history of loss of control eating

SUMMARY:
This study will investigate neural activation patterns in emotion- and cognition-related brain regions during an emotion regulation task involving cognitive reappraisal, and their associations with age and pubertal status, among overweight children and adolescents with loss of control eating as compared to overweight and normal-weight controls.

DETAILED DESCRIPTION:
Loss of control (LOC) while eating (i.e., the sense that one cannot control what or how much one is eating) is prevalent among children and adolescents. LOC eating is associated with a range of physical and psychosocial health impairments, including obesity and the development of partial- and full-syndrome eating disorders. Early identification is thus critical for preventing or minimizing these adverse health outcomes. However, little is known about the development of LOC eating in children and, consequently, there is a paucity of effective interventions. Impairments in emotion regulation appear to be involved in the onset and maintenance of eating pathology in obese samples. To date, emotion regulation in youth with LOC eating problems is poorly understood, and research on underlying neurodevelopmental substrates is virtually nonexistent. The proposed research aims to characterize neurocircuitry involved in emotion regulation among 30 overweight children with LOC eating as compared to 30 overweight and 15 normal-weight controls without LOC. Participants will complete a cognitive reappraisal task whilst situated in an MRI scanner, the purpose of which is to characterize neural activity involved in reappraisal versus an emotion maintenance control condition. The proposed research aims to advance the field's understanding of the nature and correlates of LOC eating in overweight children so as to inform intervention development.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed, aged 10-17 years.

Exclusion Criteria:

Participants will be excluded if they

* are currently taking any medications known to affect mood or weight (e.g., antidepressants, steroids);
* have a current diagnosis of a mood disorder or an eating disorder involving purging or suppressed body weight (e.g., bulimia nervosa or anorexia nervosa);
* are unable to read and understand English fluently;
* are currently pregnant;
* are a current smoker; or
* have metallic foreign bodies, face or neck tattoos, or other conditions that would prohibit fMRI scanning. Participants will complete a mock scan (see below) to ensure that their head and trunk size can be comfortably accommodated in the scanner.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 75 right-handed age- and gender-matched youth, aged 10-17 years
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Patterns of activation in cognitive control and emotion-related regions of the brain | Baseline
  Activity in cognitive control regions of the brain (i.e., dorsal anterior cingulate cortex, and dorsolateral, dorsomedial, and ventrolateral prefrontal cortices) and emotion-related regions of the brain (i.e., amygdala, insula, and ventral striatum) during emotion regulation relative to emotion maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Goldschmidt, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided